CLINICAL TRIAL: NCT07270484
Title: Rehabilitation Based on Hybrid Neuroprosthesis: Evaluation of the Feasibility, Functionality and Usability of the System in a Post-stroke Patient Population.
Brief Title: Rehabilitation Based on Hybrid Neuroprosthesis
Acronym: ReHyb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villa Beretta Rehabilitation Center (Other)
Collaborators: Technical University of Munich (Other); Össur Iceland ehf (Industry); Imperial College London (Other); Technical University of Denmark (Other); Schoen Clinic Bad Aibling (Other); Radboud University, The Netherlands (Unknown); Scuola Superiore Sant'Anna di Pisa (Other); IUVO S.r.l. (Industry); Tecnalia (Unknown)
Responsible Party: Principal Investigator, Dr. Franco Molteni, Medical Doctor, Villa Beretta Rehabilitation Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 871767
Record Dates: First submitted 2025-09-12; First posted 2025-12-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Post Stroke
Keywords: post stroke; Rehabilitation; Robobotics; Hybrid; Exoskeleton

STUDY DESIGN:
Intervention Model Description: 6 patients per platform in each clinical site were enrolled. This led to a total sample size of 24 patients. The 24 patients defined as the sample size was considered appropriate for feasibility evaluation since the system was composed by two different platforms related to the different needs patients may have according to their clinical conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehyb Device: High-Powered Platform (Experimental): Patients with lower residual mobility were assigned to the High-Powered platform (ReHyb-HPP).
  Patients assigned to ReHyb-HPP received upper limb mobilization, with active assistance, and Functional Electrical Stimulation.
  Interventions: Device: ReHyb-HPP
- ReHyb Device: Low-Powered Platform (Experimental): Patients with higher residual mobility were assigned to the Low-Powered platform (ReHyb-LPP). Patients assigned to ReHyb-LPP received upper limb mobilization, with passive assistance, and Functional Electrical Stimulation.
  Interventions: Device: ReHyb-LPP

INTERVENTIONS:
Device: ReHyb-HPP — Up to 7 sessions lasting approximately 60 minutes will be carried out, including dressing and undressing the exoskeleton and/or electrodes. At the end of the third and fifth training sessions, some questionnaires will be administered.
  At the end of each training session, the patient's adherence to the selected platform configuration will be reassessed and modified as appropriate to ensure the subject's comfort and, at the same time, to evaluate the platform's adaptability to the subject's specific conditions.
  Together with Functional electrical stimulation, patients received active assistance during predefined repetitive movements of the upper limb playing a single game.
  Arms: Rehyb Device: High-Powered Platform
Device: ReHyb-LPP — Up to 7 sessions lasting approximately 60 minutes will be carried out, including dressing and undressing the exoskeleton and/or electrodes. At the end of the third and fifth training sessions, some questionnaires will be administered.
  At the end of each training session, the patient's adherence to the selected platform configuration will be reassessed and modified as appropriate to ensure the subject's comfort and, at the same time, to evaluate the platform's adaptability to the subject's specific conditions.
  Together with Functional electrical stimulation, patients received passive assistance only at the shoulder level, during unstructured movements of the upper limb playing games with adaptive difficulty.
  Arms: ReHyb Device: Low-Powered Platform

SUMMARY:
The study is a pilot, multi-center, prospective, and open study to test feasibility, functionality and usability of a device defined as a hybrid neuroprosthesis.

DETAILED DESCRIPTION:
The ReHyb project, being oriented towards the development of a hybrid, modular, flexible and patient-specific upper-body hybrid neuro-prosthesis, potentially able to maximize the training efficacy during hospital stay as well as home-based rehabilitation or assistance during Activities of Daily Living (ADL), offering at the same time a pleasant user experience, has led to the development and integration of different modules in an attempt to adapt to the specific conditions of different patients. This goal has oriented the Consortium toward a participatory design (PD) and an ethics-by-design approach (EbD) that has been applied all along the execution of the project.

Under this perspective, two platforms have been developed and evaluated according to the following:

- Evaluation of platforms: The global evaluation of the ReHyb system and its two developed platforms, High Power Platform (HPP) and Low Power Platform (LPP). To meet this goal, a pilot, multicenter, prospective, and open study was defined to test feasibility, functionality and usability of the two platforms that constitute the hybrid neuro-prosthesis developed. A total of 24 post-stroke patients (12 per clinical site) were recruited during a time-span of 12 months for the evaluation of the ReHyb system. This number was considered sufficient for the statistical analysis to investigate the feasibility and usability of the platforms. Furthermore, the sample size is expected to allow for finding most of the usability problems.

When evaluating the ReHyb platforms in full and in their different module combinations, the ReHyb project has incorporated two different hardware devices: a stationary high powered device (ReHyb-HP) and a portable spring-loaded device (ReHyb-SL), which are both integrated with FES support. The software components include the control algorithms of the platforms, a training environment (e.g., the Rehabilitations Gaming System (RGS), a desktop Virtual Reality (VR) setup with gamified protocols for motor and cognitive rehabilitation), and the Digital Twin (e.g., the level of task difficulty and the amount of support will be adapted to the capabilities of the user).

The general scope of the studies herein presented is about evaluating the developed ReHyb System regarding its feasibility, functionality and usability rather than about evaluating any therapeutic effect of using the device. As a consequence, with a maximum duration of 3 weeks and five sessions of training per subject, the study participation is probably not long enough to expect therapeutic effects induced by the hybrid training. In fact, in previous studies, a minimum of four to seven weeks of intervention was required to detect significant clinical improvements in upper limb functions.

The applied clinical investigation protocol (CIP) was the same for the two clinical rehabilitation centres namely: Schön Klinik (SK) and VALDUCE. Nevertheless, some minimal differences were registered between the two centres without major impact on the results obtained, but with interesting complementary information coming from some of the main stakeholders on the use of the new integrated devices. In particular, SK has included the evaluation made by healthcare operators and caregivers, who have been considered the closest stakeholders to patients involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (women or men aged ≥ 18 years)
* with a diagnosis of stroke either hemorrhagic or ischemic
* with a hemiparesis of the upper limb (0 ≤ MRC ≤ 4)
* in sub-acute (up to six months after acute event) or chronic condition (more than 6 months from the acute event).
* Able to sit upright for the duration of the test.
* Subjects with a level of cognitive capacity that enables him/her to follow the instructions related to the performance of exercises.

Exclusion Criteria:

* Subjects with a high level of spasticity (Modified Ashworth Scale: In general >3 except for motorized joints which may be >2)
* Pain in the affected upper limb (Numeric Rating Scale > 4)
* Severe psychiatric disorder
* Permanent neurological symptoms present immediately before stroke
* Physical conditions that can alter normal biomechanics (e.g., recent sprains or injuries, etc.)
* Pregnant or nursing women
* No written informed consent from the patient or the legal representative
* Active implantable devices (e.g., pacemaker)
* Unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Feasibility score | Day3 and Day5
  Feasibility score is assessed by means of Unified Theory of Acceptance and Use of Technology questionnaire (UTAUT, 1-7on a likert scale per each item),
Usability | Day 6
  Perceived Usability of the device from the patients perspective. Assessed with System Usability Scale (SUS) scale questionnaire. The scale ranges from 0-100.
Number of adverse Events | from enrollment to end of treatment (up to 2 weeks).
  Safety of the delivered treatment is assessed monitoring the number of Adverse Event (AE). The metric is the number of events.
Usability | Throughout the delivered treatment (up to 2 weeks).
  Usability is assessed with donning and doffing time (measured in minutes).
Feasibility score | Day 3 and Day 5
  Feasibility score of the treatment is assessed through Intrinsic Motivation Inventory (IMI, 1-7 on a likert scale per each item)
Usability | Day 3 and Day 5
  Usability from the patient's perspective i evaluated with the Flow State Scale (FSS, 1-7 on a likert scale per each item)
Feasibiliy | Day 3 and Day 5
  Feasibiliy is evaluated with the User Experience Questionnaire (UEQ, -3 to 3 on a likert scale per each item) - short.
Usability | Day 6
  Perceived physical and cognitive fatigue were assessed with NASA-Task Load index (NASA-TLX). The scale ranges from 0-100.
Usability | Day 6
  Patient satisfaction with the device was assessed with Outcome of Prosthesis Use Survey (OPUS). The scale ranges from 0-100.

SECONDARY OUTCOMES:
Assistive Torques | From enrollment to the end of treatment (up to two weeks)
  Functionality of the platform is assessed with performance of the designed assistive algorithms, and their correct functioning, namely average torques provided (measured in Nm) across sessions.
Assistance Stimulation currents | Throughout the delivered therapy (up to two weeks).
  Functionality of the platform is assessed with performance of the designed assistive algorithms, and their correct functioning, namely , average stimulation currents (measured in mA) across session.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Molteni, Medical Doctor, Principal Investigator — Villa Beretta Rehabilitation Center; Klaus Jahn, Medical Doctor, Principal Investigator — Schon Klinik Bad Aibling
Locations (2):
- Schon Klinik, Bad Aibling, Germany
- Villa Beretta Rehabilitation Center, Costa Masnaga, Lecco, Italy